CLINICAL TRIAL: NCT03206190
Title: Studying the Prodromal and Early Phase of Hereditary Spastic Paraplegia Type 4 (SPG4)
Brief Title: The preSPG4 Study - Studying the Prodromal and Early Phase of SPG4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Prinicipal Investigator, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: preSPG4
Record Dates: First submitted 2017-06-21; First posted 2017-07-02 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hereditary Spastic Paraplegia; Hereditary, Spastic Paraplegia, Autosomal Dominant
Keywords: SPG4; presymptomatic; at risk; mutation carriers; biomarkers; longitudinal progression
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two Arms are blinded (mutation carriers vs. non mutation carriers) the third arm is an open-arm for presymptomatic tested mutation carriers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mutation carrier (Experimental): The participants will be tested genetically if they carry a disease causing mutation or not. Depending on their genetic test result they will at the end of the study divided into two groups. The clinician will be blinded throughout the entire study to the genetic results.
  Interventions: Other: SPRS Score and clinical signs; Behavioral: Cognition Testing using CANTAB; Diagnostic Test: Lumbar Puncture and blood draw; Diagnostic Test: MRI; Diagnostic Test: Electrophysiology; Diagnostic Test: Testing functional performance; Diagnostic Test: Non motor symptoms
- Non-mutation carrier (Experimental): The participants will be tested genetically if they carry a disease causing mutation or not. Depending on their genetic test result they will at the end of the study divided into two groups. The clinician will be blinded throughout the entire study to the genetic results.
  Interventions: Other: SPRS Score and clinical signs; Behavioral: Cognition Testing using CANTAB; Diagnostic Test: Lumbar Puncture and blood draw; Diagnostic Test: MRI; Diagnostic Test: Electrophysiology; Diagnostic Test: Testing functional performance; Diagnostic Test: Non motor symptoms
- Known-mutation carriers but presymptomatic (Experimental): In a third arm (open arm) we will also include positive predictive tested participants which know that they are carrying a known mutation but are at inclusion into the study asymptomatic (according to the inclusion / exclusion criteria).
  Interventions: Other: SPRS Score and clinical signs; Behavioral: Cognition Testing using CANTAB; Diagnostic Test: Lumbar Puncture and blood draw; Diagnostic Test: MRI; Diagnostic Test: Electrophysiology; Diagnostic Test: Testing functional performance; Diagnostic Test: Non motor symptoms

INTERVENTIONS:
Other: SPRS Score and clinical signs — Patients will clinically characterized by using the SPRS Score and the inventory V3
Behavioral: Cognition Testing using CANTAB — Patients will be tested using the CANTAB
Diagnostic Test: Lumbar Puncture and blood draw — Biomaterial will be collected (not obligate) to compare e.g. Nfl levels in serum and CSF
Diagnostic Test: MRI — MRI will be used to reveal presymptomatic brain morphology changes (not obligate)
Diagnostic Test: Electrophysiology — Electrophysiological tests will be used to characterize patients better.
Diagnostic Test: Testing functional performance — By using the 3 minute walk, 5 stair-climb test, and 10m walking test we will try to identify and measure subclinical progression prior to disease onset
Diagnostic Test: Non motor symptoms — By using a number of different tests we try to identify other non-motor symptoms which might manifest prior to disease onset.

SUMMARY:
Study goals

1. Prospective longitudinal data on progression in the natural course of SPG4 in presymptomatic mutation carriers prior to clinical disease onset and in early stages of disease
2. Biomarkers providing objective measures of disease activity

ELIGIBILITY:
Inclusion Criteria:

* First degree relatives (parents, offspring, and sibs) of SPG4 patients or symptomatic individuals with known SPAST mutation
* Age 18 to 70 years
* Written, informed consent (patient)

Exclusion Criteria:

* No known SPAST-mutation within the family
* Manifest spastic gait (subclinical signs like increased deep tendon reflexes, positive Babinski sign are allowed)
* Participation in interventional trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Identification of a change of recognizable signs or symptoms | every two years, up to eight years
  Identification of recognizable signs or symptoms and their time course prior to disease-onset defined by the presence of a spastic gait and at least one of three additional features:
  1. manifest spasticity in the clinical examination (Ashworth Scale >0)
  2. positive Babinski sign
  3. pyramidal pattern of muscle weakness (e.g. hip abduction or foot elevation preferentially involved)

SECONDARY OUTCOMES:
Subclinical progression (10m walking time) | every two years, up to eight years
  To identify measures of subclinical progression of motor symptoms prior to disease onset by comparing functional performance in mutation carriers with that in individuals without mutation.
Subclinical progression (5-stair climbing test time) | every two years, up to eight years
  To identify measures of subclinical progression of motor symptoms prior to disease onset by comparing functional performance in mutation carriers with that in individuals without mutation.
Subclinical progression (3 minute walking test (3MW)) | every two years, up to eight years
  To identify measures of subclinical progression of motor symptoms prior to disease onset by comparing functional performance in mutation carriers with that in individuals without mutation.
MRI (not obligate) - DTI | every two years, up to eight years
  To reveal alterations in brain morphology with magnetic resonance im-aging (MRI) in presymptomatic mutation carriers by measuring diffusion tensor imaging (DTI).
MRI (not obligate) - volumetry | every two years, up to eight years
  To reveal alterations in brain morphology with magnetic resonance im-aging (MRI) in presymptomatic mutation carriers by measuring brain volumetry.
Nfl | every two years, up to eight years
  To compare Nfl levels in serum (and cerebrospinal fluid (CSF) - not obligate) in mutation carriers and non-carriers.
Non-motor symptoms (SPRS inventory V3) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the SPRS inventory V3.
Non-motor symptoms (quality of life) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the EQ-5D.
Non-motor symptoms (fatigue) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the MFI.
Non-motor symptoms (pain) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the Brief Pain Inventory.
Non-motor symptoms (depression) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the Becks Depression Inventory (BDI).
Non-motor symptoms (restless-legs) | every two years, up to eight years
  To identify clinical signs (other than spasticity) that are more frequent in mutation carriers than in non-carriers as recorded by the restless-legs diagnostic criteria questions.
SPRS | every two years, up to eight years
  To determine the sensitivity of the Spastic Paraplegia Rating Scale (SPRS) to detect the manifestation of disease onset as defined above.
Cognition (CANTAB) | every two years, up to eight years
  To compare cognitive performance by using the CANTAB battery in mutation and non-mutation carriers
Cognition (MoCA) | every two years, up to eight years
  To compare cognitive performance by using the Montreal Cognitive Assessment (MoCA) in mutation and non-mutation carriers

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Schöls, Prof., Principal Investigator — Head of Department
Locations (1):
- University Hospital Tübingen, Center for Neurology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rattay TW, Volker M, Rautenberg M, Kessler C, Wurster I, Winter N, Haack TB, Lindig T, Hengel H, Synofzik M, Schule R, Martus P, Schols L. The prodromal phase of hereditary spastic paraplegia type 4: the preSPG4 cohort study. Brain. 2023 Mar 1;146(3):1093-1102. doi: 10.1093/brain/awac155. PMID 35472722